CLINICAL TRIAL: NCT03234569
Title: Safety and Efficacy of Sonohysterosalpingography for the Evaluation of Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Pellerito, Vice Chair, Education Department of Radiology, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-0967
Record Dates: First submitted 2017-07-28; First posted 2017-07-31 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Infertility, Female
Keywords: sonohysterosalpingography; hysterosalpingography
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sonoHSG (Experimental): This is the research procedure and it will be added onto the standard of care procedure for all subjects.
  Interventions: Procedure: sonoHSG

INTERVENTIONS:
Procedure: sonoHSG — This procedure uses agitated saline to produce air bubbles at the time of the Sonohysterogram which optimizes fallopian tube visualization. The sonoHSG is free of radiation and use of contrast. In this study, in order to produce the air bubbles at the time of the sonohysterogram, the investigators will be using a continuous saline-air device that may produce a technically superior image. For the ultrasound images, General Electric will be supporting us by providing us the Voluson E10 and RIC5-9-D.

SUMMARY:
This pilot study is a collaborative effort between Northwell Health's Departments of Fertility and Radiology.The aim of this study is to evaluate the feasibility of the Sonohysterosalpingography (sonoHSG) for it to be determined as the standard of care. Additionally, it aims to improve the work up of infertility by integrating the examination of structural abnormalities of the Fallopian tubes and uterus into a single radiation free ultrasound guided procedure, the sonoHSG.

DETAILED DESCRIPTION:
This pilot study is a collaborative effort between Northwell Health Fertility and the Radiology Department to streamline the fertility evaluation process and reduce the burden of stress many fertility patients experience by eliminating an imaging examination which is painful and exposes the patient to potentially harmful radiation.

The aim of this study is to improve the workup of infertility by integrating the examination of structural abnormalities of the fallopian tubes and uterus into a single radiation-free ultrasound guided procedure, the sonohysterosalpingogram (sonoHSG). Confirmation of tubal patency is extremely important as approximately 25-35% of female infertility can be attributed to fallopian tube pathology. The current paradigm is to use two separate imaging exams; the hysterosalpingogram (HSG), a transvaginal procedure that uses radiation and iodinated contrast to visualize the fallopian tubes, and the sonohysterogram, a transvaginal procedure that uses ultrasound and saline to visualize the uterus. By using agitated saline, to produce air bubbles, fallopian tube visualization is optimized during the time of sonohysterogram (sonoHSG). The investigators plan to also utilize a continuous saline-air device that may produce a technically superior sonoHSG.

As a result of this study, the Radiology Department and Northwell Health Fertility will work together to encourage, educate, and support physicians to promote the utility of sonoHSG as the first imaging examination for the infertility workup. Currently, this institution is not routinely utilizing the sonoHSG despite the advantages in safety, comfort, and convenience to the patient. The investigators aim to effect a change in the current practice at this institution by increasing the knowledge and visibility of the sonoHSG by creating educational materials for referring physicians, and creating a pilot program that demonstrates the value and efficacy of the exam. SonoHSG can be performed concurrently at the time of the sonohysterogram at no additional cost to the patient.

The investigators will enroll 30 patients from Northwell Health Fertility over the course of one year. Measures of success will include concordance between sonoHSG and HSG in patients who receive both procedures, and patient surveys evaluating pain utilizing the pain scale. If sonoHSG proves to be efficacious, future steps will be to educate referring physicians and patients about the utility of the examination using print materials and a grand rounds lecture. The investigators will also measure the number of sonoHSGs ordered compared to HSGs for the evaluation of fallopian tube patency in order to evaluate if there has been a shift in the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing evaluation for infertility in the Northwell Health System
* Non-pregnant women age 18-50 years old
* Subject is not menstruating at the time of study
* Provide written informed consent and written HIPAA authorization prior to study initiation
* Willing to comply with the specified follow-up evaluation schedule

Exclusion Criteria:

* History of active pelvic infection
* History of tubal ligation or salpingectomy
* History of adverse reaction to iodinated contrast
* Subject is pregnant
* Subject is menstruating at time of study
* Subject is unable to participate in study evaluations pre- and post-treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Concordance between sonoHSG and HSG results. The sonoHSG and HSG will be considered interchangeable if the level of agreement between them is >= 80%. | 1 year

SECONDARY OUTCOMES:
Quantification of level of patient pain in regard to sonoHSG versus HSG | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Pellerito, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maheux-Lacroix S, Boutin A, Moore L, Bergeron ME, Bujold E, Laberge PY, Lemyre M, Dodin S. Hysterosalpingosonography for diagnosing tubal occlusion in subfertile women: a systematic review protocol. Syst Rev. 2013 Jul 4;2:50. doi: 10.1186/2046-4053-2-50. PMID 23826862
- [Background] Exacoustos C, Zupi E, Carusotti C, Lanzi G, Marconi D, Arduini D. Hysterosalpingo-contrast sonography compared with hysterosalpingography and laparoscopic dye pertubation to evaluate tubal patency. J Am Assoc Gynecol Laparosc. 2003 Aug;10(3):367-72. doi: 10.1016/s1074-3804(05)60264-2. PMID 14567814
- [Background] Marci R, Marcucci I, Marcucci AA, Pacini N, Salacone P, Sebastianelli A, Caponecchia L, Lo Monte G, Rago R. Hysterosalpingocontrast sonography (HyCoSy): evaluation of the pain perception, side effects and complications. BMC Med Imaging. 2013 Aug 23;13:28. doi: 10.1186/1471-2342-13-28. PMID 23968513
- [Background] Luciano DE, Exacoustos C, Luciano AA. Contrast ultrasonography for tubal patency. J Minim Invasive Gynecol. 2014 Nov-Dec;21(6):994-8. doi: 10.1016/j.jmig.2014.05.017. Epub 2014 Jun 6. PMID 24910933
- [Background] Schankath AC, Fasching N, Urech-Ruh C, Hohl MK, Kubik-Huch RA. Hysterosalpingography in the workup of female infertility: indications, technique and diagnostic findings. Insights Imaging. 2012 Oct;3(5):475-83. doi: 10.1007/s13244-012-0183-y. Epub 2012 Jul 17. PMID 22802083
- [Background] Szymusik I, Grzechocinska B, Marianowski P, Kaczynski B, Wielgos M. Factors influencing the severity of pain during hysterosalpingography. Int J Gynaecol Obstet. 2015 May;129(2):118-22. doi: 10.1016/j.ijgo.2014.11.015. Epub 2015 Jan 27. PMID 25650318
- [Background] Handelzalts JE, Levy S, Peled Y, Binyamin L, Wiznitzer A, Goldzweig G, Krissi H. Information seeking and perceptions of anxiety and pain among women undergoing hysterosalpingography. Eur J Obstet Gynecol Reprod Biol. 2016 Jul;202:41-4. doi: 10.1016/j.ejogrb.2016.04.037. Epub 2016 Apr 30. PMID 27160813
- See also: Sonohysterosalpingography: A suitable choice in infertility work up — https://link.springer.com/content/pdf/10.1007/s10396-012-0417-0.pdf

DOCUMENTS (2):
  • Study Protocol (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03234569/Prot_000.pdf
  • Informed Consent Form (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03234569/ICF_001.pdf